CLINICAL TRIAL: NCT06778356
Title: Effect of Environment on the Central and Peripheral Nervous System
Acronym: RUMI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Susan Rodriguez, PhD student, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY007343
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Rumination
Keywords: Rumination, nature exposure, respiratory sinus arrhythmia, blood pressure
MeSH Terms: conditions — Rumination Syndrome; Arrhythmia, Sinus | interventions — Built Environment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Built environment assignment (Experimental): Participants will complete the study session in a built environment
  Interventions: Other: Built environment
- Natural environment (Experimental): Participants will complete the study session in a natural environment.
  Interventions: Other: Natural environment

INTERVENTIONS:
Other: Built environment — Participants will complete the study session at a University student center.
  Arms: Built environment assignment
Other: Natural environment — Participants will complete the study session in a nature trail.
  Arms: Natural environment

SUMMARY:
The main goal of this study is to understand how different environments influence both mental responses, like overthinking (rumination), and physical reactions, such as heart rate and blood pressure, after a challenging task.

DETAILED DESCRIPTION:
This study aims to explore the restorative effects of nature exposure on rumination- a mental process that affects attention-and cardiovascular responses to a challenging task. A total of 95 participants will be randomly assigned to either a built or natural environment. Each participant will take part in a 2.5-hour session. Initially, an electrocardiogram (ECG) will be attached to measure heart activity. Participants will then engage in a 30-minute task designed to immerse them in their assigned environment (the ABC engagement task). Following this, they will have a 10-minute period of quiet relaxation to establish baseline cardiovascular measures. After baseline, participants will complete a challenging task (the Remote Associates Test (RAT)), which is designed to induce sympathetic arousal. Afterward, they will rest quietly for another 10 minutes to monitor cardiovascular recovery. Finally, participants will complete post-task surveys through Qualtrics, assessing their state of rumination, perceived difficulty of the task, effort levels, and expectations of success.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18 years of age or older.

Exclusion Criteria:

* Individuals with a history of cardiovascular disease or disorders, those who are pregnant, or are taking medications which may alter/affect cardiovascular function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
Respiratory Sinus Arrhythmia (RSA) | Respiratory sinus arrhythmia will be measured during a baseline (20 minutes), challenging task (19 minutes) and the recovery period (10 minutes).
Blood pressure | Systolic (SBP) and diastolic blood pressure (DBP) will be measured during a baseline (20 minutes), challenging task (19 minutes), and recovery period (10 minutes).
Remote Associates Test (RAT) | Participants will complete the RAT task for 19 minutes (44 trials).
  In this study, the remote associates test (RAT) will be used as a challenging task to induce sympathetic arousal. Each RAT item consists of three words, participants will be asked to generate a fourth word/solution associated with the words presented by means of a compound word, synonymy, or semantic association. The participant has provided a fourth/solution word or the 30 second time limit. The task will consist of a total of 39 trials, including 5 practice trials.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No